CLINICAL TRIAL: NCT02913573
Title: Pectoral Nerve Block vs. Standard Anesthesia in Patients Undergoing Mastectomy and Immediate Breast Reconstruction: Impact on Post-operative Pain and Nausea/Vomiting
Brief Title: Effect of Pectoral Nerve Block on Post-op Pain in Patients Undergoing Mastectomy and Immediate Reconstruction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huntington Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jeannie Shen, Director, Breast Surgery, Huntington Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31801/1
Record Dates: First submitted 2016-09-19; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GA + Pec Block (Experimental): Following induction of general anesthesia, the patients in the intervention group will undergo an ultrasound-guided pectoral block. With the patient in proper position, the infraclavicular and axillary regions are prepped with chlorhexidine. An US probe is placed below the third of the clavicle over the pectoralis major muscle. After identifying the appropriate anatomical structures, a 21-gauge echogenic needle is advanced under US visualization to the tissue plane between the pectoral major and pectoral minor muscles where the lateral and medial pectoralis nerves lie and 15 mL of 0.25% bupivacaine will be deposited. In a similar manner, 20 mL of 0.25% bupivacaine will be deposited under ultrasound-guidance at the level of the third rib above the serratus anterior muscle.
  Interventions: Device: Ultrasound; Drug: 0.25% bupivacaine
- GA only (No Intervention): Patients will receive standard general anesthesia.

INTERVENTIONS:
Device: Ultrasound — Pectoral nerve block is a regional block administered under ultrasound guidance which blocks the nerves of the thorax and chest areas.
  Arms: GA + Pec Block
Drug: 0.25% bupivacaine — Pectoral nerve block is a regional block administered under ultrasound guidance where 15 mL of 0.25% bupivacaine is instilled between the pectoral major and pectoral minor muscles where the lateral and medial pectoralis nerves lie. In a similar manner, 20 mL of 0.25% bupivacaine will be deposited under ultrasound-guidance at the level of the third rib above the serratus anterior muscle.
  Other Names: 0.25% Marcaine
  Arms: GA + Pec Block

SUMMARY:
Patients undergoing total mastectomy with immediate breast reconstruction with a tissue expander or implant under general anesthesia will be randomly assigned to the addition of a pectoral nerve block or no regional block. Post-operative pain, nausea/vomiting scores will be assessed.

DETAILED DESCRIPTION:
Patients undergoing total mastectomy with immediate breast reconstruction with a tissue expander or implant under general anesthesia will be randomly assigned to the addition of a pectoral nerve block or no regional block after induction of general anesthesia and prior to the start of surgery. Post-operative pain scores and post-operative pain medication usage will be recorded. Post-operative nausea/vomiting scores and post-op anti-emetic medication usage will be recorded. The clinical impact of pectoral nerve block on this expanding population of patients will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18-90 years old
2. Subjects able to read and understand the informed consent
3. American Society of Anesthesiologists (ASA) physical status I and II
4. Subjects scheduled to undergo unilateral or bilateral mastectomy with immediate breast reconstruction with submuscular placement of tissue expander or permanent implant under general anesthesia, including:

   * subjects diagnosed with breast cancer
   * subjects diagnosed with atypia or other high risk proliferative breast disease
   * subjects with a family history who are considered at high risk for breast cancer (including those with hereditary or genetic predisposition)

Exclusion Criteria:

1. Subjects unable to read or understand the informed consent
2. ASA physical status III or IV
3. Subjects with an allergy to local anesthetic
4. Subjects with a medical contraindication to regional anesthetic, such as coagulopathy or local infection
5. Subjects with a pre-existing submuscular implant
6. Subjects scheduled to undergo mastectomy with myocutaneous flap reconstruction
7. Subjects scheduled to undergo mastectomy without immediate reconstruction
8. Subjects with a history of chronic pain or chronic opioid use

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Post-op pain | within first 48 hours
  post-op pain assessed by Visual Analog Scale

SECONDARY OUTCOMES:
Post-op nausea/vomiting | within first 48 hours
  post-op nausea/vomiting score assessed on standard scale

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie Shen, MD, Principal Investigator — Huntington Memorial Hospital
Locations (1):
- Huntington Memorial Hospital, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Result] Leiman D, Barlow M, Carpin K, Pina EM, Casso D. Medial and lateral pectoral nerve block with liposomal bupivacaine for the management of postsurgical pain after submuscular breast augmentation. Plast Reconstr Surg Glob Open. 2015 Jan 8;2(12):e282. doi: 10.1097/GOX.0000000000000253. eCollection 2014 Dec. PMID 25587516
- [Result] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Result] Wu J, Buggy D, Fleischmann E, Parra-Sanchez I, Treschan T, Kurz A, Mascha EJ, Sessler DI. Thoracic paravertebral regional anesthesia improves analgesia after breast cancer surgery: a randomized controlled multicentre clinical trial. Can J Anaesth. 2015 Mar;62(3):241-51. doi: 10.1007/s12630-014-0285-8. Epub 2014 Dec 6. PMID 25480319
- [Result] Pei L, Zhou Y, Tan G, Mao F, Yang D, Guan J, Lin Y, Wang X, Zhang Y, Zhang X, Shen S, Xu Z, Sun Q, Huang Y; Outcomes Research Consortium. Ultrasound-Assisted Thoracic Paravertebral Block Reduces Intraoperative Opioid Requirement and Improves Analgesia after Breast Cancer Surgery: A Randomized, Controlled, Single-Center Trial. PLoS One. 2015 Nov 20;10(11):e0142249. doi: 10.1371/journal.pone.0142249. eCollection 2015. PMID 26588217
- [Result] Fahy AS, Jakub JW, Dy BM, Eldin NS, Harmsen S, Sviggum H, Boughey JC. Paravertebral blocks in patients undergoing mastectomy with or without immediate reconstruction provides improved pain control and decreased postoperative nausea and vomiting. Ann Surg Oncol. 2014 Oct;21(10):3284-9. doi: 10.1245/s10434-014-3923-z. Epub 2014 Jul 18. PMID 25034821
- [Result] Byrne K, Levins KJ, Buggy DJ. Can anesthetic-analgesic technique during primary cancer surgery affect recurrence or metastasis? Can J Anaesth. 2016 Feb;63(2):184-92. doi: 10.1007/s12630-015-0523-8. PMID 26497721
- [Result] Cassinello F, Prieto I, del Olmo M, Rivas S, Strichartz GR. Cancer surgery: how may anesthesia influence outcome? J Clin Anesth. 2015 May;27(3):262-72. doi: 10.1016/j.jclinane.2015.02.007. Epub 2015 Mar 11. PMID 25769963